CLINICAL TRIAL: NCT00237536
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Comparison Study of the Efficacy and Safety of Lonidamine for the Treatment of Symptomatic Benign Prostatic Hyperplasia
Brief Title: Study of the Efficacy and Safety of Lonidamine for the Treatment of Symptomatic Benign Prostatic Hyperplasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Threshold Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TH-CR-203
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; BPH; Enlarged Prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — lonidamine

INTERVENTIONS:
Drug: Lonidamine

SUMMARY:
The purpose of this trial is to evaluate the dose response relationship of lonidamine and the primary efficacy endpoint, International Prostate Symptom Score (IPSS), in subjects with symptomatic benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the purpose and risks of the study and sign a statement of informed consent
2. Male 65-80 years of age (or 40-80 with vasectomy). Vasectomized men must have documentation of azoospermia.
3. Presence of LUTS (lower urinary tract symptoms) for at least 3 months
4. Prostate volume measured by TRUS (transrectal ultrasound) > 30 cc
5. Qmax < 15 mL/sec when measured by uroflowmetry (minimum of 125 mL must be voided)
6. IPSS (International Prostate Symptom Score) > 12
7. PSA > 1.0 ng/mL
8. Must ensure and consent to use medically acceptable methods of contraception throughout the entire study with sexual partners of childbearing potential
9. Able to comply with the prescribed treatment protocol and evaluations

Exclusion Criteria:

1. Prior treatment for BPH with alpha blockers and/or herbal supplements for the treatment of BPH in the past 2 weeks (alpha-blockers and/or herbal supplements for the treatment of BPH are not allowed during the study). Prior treatment with 5-alpha reductase inhibitors is allowed if discontinued at least 3 months prior to enrollment.
2. Prior surgery of the prostate (except biopsies; subject is eligible to enroll one month after full recovery from prostate biopsy.)
3. Current or past evidence of malignant disease of the prostate or prostatic intraepithelial neoplasia (For subjects with PSA between 4 - 10 ng/mL, prostate cancer must be ruled out to the satisfaction of the Principal Investigator. Subjects with PSA >10 ng/mL are excluded).
4. Active urinary tract infections (UTI)
5. Active cardiac, renal or hepatic disease as evidenced by:

   1. Serum creatinine > 1.8 mg/dL
   2. ALT or AST > 2.5x the upper limit of normal
   3. History of active myocardial infarction, unstable cardiac arrhythmias, or stroke within 6 months prior to screening
   4. Uncontrolled congestive heart failure
6. Uncontrolled diabetes mellitus (fasting blood glucose > 200 mg/dL)
7. Use of systemic steroids for any reason (systemic steroid usage is not allowed during the study). Inhaled and/or topical steroids are allowed.
8. Concurrent participation or participation in an investigational drug study within the past 30 days prior to screening
9. Concomitant disease or condition that could interfere with the conduct of the study, or would in the opinion of the Investigator, pose an unacceptable risk to the subject

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240
Dates: Start 2005-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
IPSS

SECONDARY OUTCOMES:
Maximum urinary flow rate (Qmax)
Post-void residual urine volume (PVR)
Prostate volume
Prostate specific antigen (PSA)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - Chris B. Threatt, MD Inc., Atherton, California
  - Urological Sciences Research Foundation, Culver City, California
  - Atlantic Urological Medical Group, Long Beach, California
  - California Professional Research, Newport Beach, California
  - San Diego Uro-Research, San Diego, California
  - Stanford University Hospital, Stanford, California
  - Urology Research Options, Aurora, Colorado
  - Connecticut Clinical Research Center Urology Specialists, Waterbury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Florida Healthcare Research, Ocala, Florida
  - Midwest Prostate & Urology Health Center, Chicago, Illinois
  - Specialty Care Research, Peoria, Illinois
  - Northeast Indiana research, LLC, Fort Wayne, Indiana
  - Metropolitan Urology, Jeffersonville, Indiana
  - Werner, Murdock & Francis, PA, Urology Associates, Greenbelt, Maryland
  - Sheldon J. Freedman, MD Ltd., Las Vegas, Nevada
  - Delaware Valley Clinical Research, Cherry Hill, New Jersey
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Urology Healthcare Associates, Woodlane, New Jersey
  - Accumed Research Associates, Garden City, New York
  - New York University School of Medicine, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Radiant Research. Columbus, Columbus, Ohio
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - State College Urologic Associates, State College, Pennsylvania
  - University Urological Research Institute, Providence, Rhode Island
  - Radiant Research, Greer, Greer, South Carolina
  - UT Southwestern Medical Center at Dallas, Dept of Urology, Dallas, Texas
  - Accelovance, Houston, Texas
  - Baylor College of Medicine, Scott Department of Urology, Houston, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Integrity Medical Research, LLC, Mountlake Terrace, Washington